CLINICAL TRIAL: NCT02584270
Title: Prosthesis Guided Speech Rehabilitation of T1/T2 Cancers of the Tongue (PGSRT): a Randomized Clinical Trial
Brief Title: Prosthesis Guided Speech Rehabilitation of T1/T2 Cancers of the Tongue
Acronym: PGSRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Stephanie M. Munz, Clinical Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00093723.1
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Tongue Neoplasms; Tongue Cancer; Oral Cancer
Keywords: palatal drop prosthesis
MeSH Terms: conditions — Tongue Neoplasms; Mouth Neoplasms | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prosthesis + Articulation Therapy (Experimental): This arm will receive a PAP (palatal augmentation prosthesis) with standard articulation therapy. This is the study arm
  Interventions: Device: Palatal Augmentation Prosthesis (PAP); Other: Articulation Therapy
- No Prosthesis; Articulation Therapy Only (Other): This arm will not receive a PAP (palatal augmentation prosthesis), but will receive standard articulation therapy. This is the control arm.
  Interventions: Other: Articulation Therapy

INTERVENTIONS:
Device: Palatal Augmentation Prosthesis (PAP) — The palatal augmentation prosthesis, or PAP can improve speech and swallowing functions through reshaping the palatal contours. This may improve the contact between the tongue and hard palate as a person speaks or eats. It is meant to be created after adequate healing in patients with adequate motivation for improvements in their speech and swallowing. Regular wear and articulation therapy are necessary for this therapy to be effective.
  Arms: Prosthesis + Articulation Therapy
Other: Articulation Therapy — Subjects will receive the standard of care speech and articulation therapy in either arm.
  Other Names: Speech Therapy

SUMMARY:
This study will fill a scientific gap in the current knowledge providing data for evaluation of the palatal augmentation prosthesis (PAP) as a therapeutic modality post-surgery. This is a robust scientific randomized prospective clinical trial.

Positive outcomes from this study have the potential to dramatically alter the most common issues of oral cancer therapy, namely speech and swallowing functions. Patients will have been diagnosed with a cancer lesion of the tongue requiring surgery and removal of part of the tongue. Smaller cancers of the tongue are sized as T1 or T2. For patients with smaller lesions, a PAP, which can aid in speaking and swallowing, is not routinely provided.

DETAILED DESCRIPTION:
This study will randomize patients into two arms; one for oral cancer patients that receive a small device, similar to a denture, called a PAP. The other arm will be patients who serve as a control and will not receive a PAP.

The PAP requires patients to have a dental mold created. A dentist customizes the PAP to specifically fit the individual's mouth.

The study will investigate whether the PAP improves speech following tongue cancer as measured by three different scales. Both groups will see a speech language therapist for additional measures of speech evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new diagnosis of a T1/T2 tongue cancer

Exclusion Criteria:

* Patients with recurrent disease
* Patients with a history of prior head and neck radiation therapy
* Patients who lack adequate maxillary dentition to support a palatal augmentation prosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Word intelligibility | 6 months
  The Assessment of Intelligibility of Dysarthric speech (AIDS) test is a validated assessment of word and sentence intelligibility as well as speech efficiency. The AIDS score will be measured at baseline before surgery for tongue cancer, then after surgery at the timepoints of one month, three months, six months and one year. Six months is the primary time point measurement. Measurements will also be obtained at these other time points, which will possibly be used for other outcome analysis which are neither primary nor secondary. The unit being measured will be a percent score of words correctly transcribed by two blinded untrained listeners of the subjects' audio recordings of separate un-related words.

SECONDARY OUTCOMES:
Sentence intelligibility | 6 months
  The Assessment of intelligibility of dysarthric speech (AIDS) test is a validated assessment of word and sentence intelligibility as well as speech efficiency and will be measured at baseline before surgery for tongue cancer, then post-operatively at one month, three months, six months and one year. Six months is the primary time point measurement, although measurements will also be obtained at these other time points, which will possibly be used for other outcome analysis which are neither primary nor secondary. The unit being measured will be a percent score of words correctly transcribed by two blinded untrained listeners of the subjects' audio recordings of words in sentences.
Articulation at the word level of phonemes (consonant sounds) | 6 months
  The Goldman Fristoe 2 test of Articulation sounds in words subtest (GFTA2) is a standardized, validated and reliable tool that systematically assesses articulation of phonemes (consonant sounds). It offers normative data from ages 2 through 21. This will be measured at baseline pre-treatment of tongue cancer, then post-operatively at one month, three months, six months and one year. Six months is the primary time point measurement, although measurements will also be obtained at these other time points, which will possibly be used for other outcome analysis which are neither primary nor secondary. The unit being measured is the raw score generated from the test.
Patient satisfaction with speech | 6 months
  The Speech Handicap Index (SHI) is designed to evaluate an individual's speech function and corresponding psycho-social factors. This will be measured at baseline pre-treatment of tongue cancer, then post-operatively at one month, three months, six months and one year. Six months is the primary time point measurement, although measurements will also be obtained at these other time points, which will possibly be used for other outcome analysis which are neither primary nor secondary. The unit being measured is the mean score of the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Munz, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Department of Oral and Maxillofacial Surgery and Hospital Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No